CLINICAL TRIAL: NCT04524338
Title: Longitudinal Study Examining At-Home Transcranial Direct Current Stimulation
Brief Title: Longitudinal Study Examining At-Home tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Carlos Roncero, Consultant, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2020-1885
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At Home tDCS Users (Experimental): Participants conducting tDCS at home
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Brain Stimulation Devices attached to scalp
  Other Names: tDCS

SUMMARY:
Participants with dementia have reported improvements after receiving tDCS in a study at our lab. Although we make an effort to enroll such participants in further tDCS research studies, some participants are ineligible for further studies or simply unwilling to continue being a research participant. These same individuals, however, are interested in purchasing their own tDCS machine and have approached us for advice on how to purchase their own machine. Because these devices are commercially available, there is nothing theoretically stopping these participants from purchasing their own machine. Therefore, we have chosen to carry out a longitudinal study that will allow us to serve as an advisory role for participants who have decided to continue administering tDCS at home. We will recommend the tDCS related items that should be purchased, and train participants on how to properly administer tDCS. Monthly reports will also be collected, which will allow us to monitor the person's condition. We plan to monitor participants for at least two years. From these reports, we will be able determine to what extent tDCS is beneficial when done at home as a treatment for dementia symptoms.

DETAILED DESCRIPTION:
In the past decade, several studies have noted that the application of transcranial direct current stimulation (tDCS) when applied to the scalp of a person with dementia, as they completed a training task in a particular domain, can lead to improved performance on that task (liu, Rau, Gallagher, Rajji, Lanctot, & Hermann, 2017). In our own lab, we have also seen improvements in response to the application of TdCS. For example, we found that applying transcranial direct current stimulation (tDCS) to people with dementia led to an improvement in naming ability (Roncero, Kniefel, Service, Thiel, Probst, & Chertkow, 2017). Recently, we have initiated additional studies in domains such as executive function and memory. These studies remain in progress, but participants have again shown improvement, and the improvement is noted by the families. Some of the participants who completed a tDCS study in our lab are so impressed by the results that they have approached us about the purchase of their own tDCS machine. Some of these participants have even tried medication in the past and report tDCS is more effective. Because tDCS machines are commercially available, these individuals could in theory go about buying their own machines at their own initiative; however, participants would prefer our assistance obtaining a machine and be trained on how to administer tDCS at home.

Proposed Study We will assist participants obtain their own tDCS machine, we have decided to do so in the form of a longitudinal study. More specifically, we plan to assist participants obtain their own machine and train them on the administration of tDCS, but will also collect longitudinal data from them. We will obtain monthly reports that will allow us to monitor whether stimulation remains effective and the general condition of the participant for at least two years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's Disease or other form of dementia (e.g., Primary Progressive Aphasia)

Exclusion Criteria:

* Metal in the head or other factors that would make stimulation unsafe

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
General Cognition | two years
  Improved General Cognition as defined by scores on the Montreal Cognitive Assessment. Test has scores from 0-30, where higher scores reflect better cognition. In this study, an increased score would reflect an improvement in general cognition, which we would interpret as associated with the application of transcranial direct current stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roncero, PhD, Principal Investigator — Baycrest
Locations (1):
- Perform Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No